CLINICAL TRIAL: NCT00531908
Title: Physiopathology of Sodium Retention in Acromegaly
Acronym: AcromEnaC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P061012
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2008-08

CONDITIONS: Acromegaly
Keywords: Growth Hormone; Epithelial sodium channel; Hypertension; A Furosemide; Nasal Mucosa
MeSH Terms: conditions — Acromegaly; Hypertension | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): To compare natriuretic effect of a single dose administration of amiloride (20 mg) in patients with acromegaly
  Interventions: Drug: furosemide

INTERVENTIONS:
Drug: furosemide — furosemide

SUMMARY:
Acromegaly is a disease due to an excess of growth hormone that abnormally occurs in adulthood. It is due to a benign (non cancerous) tumor located in a particular part of the brain that secretes several hormones, the hypophysis. The excess of growth hormones in adults induces an increase in bone (resulting in large enlargement of extremities), and organs. The disease is complicated by the apparition of cardiovascular events including retention of water, salt in the tissues and increase in blood pressure, that altogether might major the mortality of the patients. The investigators recently got experimental data suggesting that the retention of water and salt is mainly due to the activation by the growth hormone of a renal transporter of sodium. Because this transporter is highly sensitive to amiloride, a well know diuretic, the investigators hypothesize that this drug will be very efficient in treating the hypertension in patients, as compared to another diuretic, furosemide.

DETAILED DESCRIPTION:
To prove this, we compared the response to amiloride administrated before and after treatment of acromegaly in the same subject. We will also compare the response to furosemide administrated before and after treatment of acromegaly in the same subject. We expected that the response to amiloride will be greater before than after treatment, while the response to furosemide will be lesser before than after treatment.

Detailed Description:

Definition: Extended description of the protocol, including information not already contained in other fields, such as comparison(s) studied.

Patients will be recruited in the Department of Endocrinology and Reproductive diseases in BICETRE University Hospital and will be explored in the Centre for Clinical Investigation of HEGP. Investigations will be performed during 4 separate day-hospital stays (2 pre-treatment and 2 post treatment) in the CIC of HEGP. The tests will consist of blood and urine sample collections before and after a single dose administration of furosemide or amiloride. The tests will be performed before treatment of acromegaly in random order and separated by 48hours, interval performed before treatment, and repeated in the same order after normalization of IGF1 by appropriate treatment.

The study will last for 2 years, with a 12 months maximal participation of each patient

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 75 yrs
* proven evolutive acromegalia with indication of treatment (surgical or medical)
* controlled blood pressure (systolic BP < 140 mmHg et diastolic BP < 90 mmHg)
* signed informed consent
* efficient contraception in women

Exclusion Criteria:

* edematous state unrelated to acromegaly
* history of sulfamide intolerance
* hemoglobin < 8g/dL
* pregnant or breastfeeding women
* inability to give informed consent
* blood donation in the preceding 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To compare natriuretic effect of a single dose administration of amiloride (20 mg) in patients with acromegaly | before and after treatment of acromegaly.

SECONDARY OUTCOMES:
To compare natriuretic effect of a single dose of furosemide (bolus 5 mg, then 10 mg over 2 hrs) in patients with acromegaly | before and after treatment of acromegaly.
To study the difference of the intranasal potential | before and after treatment of acromegaly.

CONTACTS AND LOCATIONS:
Overall Officials: Peter KAMENICKY, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Bicetre, Paris, France

REFERENCES:
- [Result] Bihan H, Espinosa C, Valdes-Socin H, Salenave S, Young J, Levasseur S, Assayag P, Beckers A, Chanson P. Long-term outcome of patients with acromegaly and congestive heart failure. J Clin Endocrinol Metab. 2004 Nov;89(11):5308-13. doi: 10.1210/jc.2004-0821. PMID 15531475
- [Derived] Kamenicky P, Blanchard A, Gauci C, Salenave S, Letierce A, Lombes M, Brailly-Tabard S, Azizi M, Prie D, Souberbielle JC, Chanson P. Pathophysiology of renal calcium handling in acromegaly: what lies behind hypercalciuria? J Clin Endocrinol Metab. 2012 Jun;97(6):2124-33. doi: 10.1210/jc.2011-3188. Epub 2012 Apr 10. PMID 22496496
- [Derived] Kamenicky P, Blanchard A, Frank M, Salenave S, Letierce A, Azizi M, Lombes M, Chanson P. Body fluid expansion in acromegaly is related to enhanced epithelial sodium channel (ENaC) activity. J Clin Endocrinol Metab. 2011 Jul;96(7):2127-35. doi: 10.1210/jc.2011-0078. Epub 2011 Apr 20. PMID 21508131